CLINICAL TRIAL: NCT00002456
Title: Postgrafting Methotrexate and Cyclosporine for the Prevention of Graft-Versus-Host Disease
Brief Title: Graft-Versus-Host Disease Prevention in Treating Patients Who Are Undergoing Bone Marrow Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Purpose: Supportive Care
Other Study IDs: 267.01; FHCRC-267.01; FHCRC-267.00; NCI-V86-0145; CDR0000074146 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-04-26 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma
Keywords: recurrent childhood acute lymphoblastic leukemia; childhood non-Hodgkin lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; recurrent adult non-Hodgkin lymphoma; graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — Cyclosporine; Methotrexate

INTERVENTIONS:
Drug: cyclosporine
Drug: methotrexate
Procedure: allogeneic bone marrow transplantation

SUMMARY:
RATIONALE: Bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy used to kill tumor cells. Sometimes the transplanted cells can make an immune response against normal tissues. Methotrexate and cyclosporine may prevent this from happening.

PURPOSE: Phase III trial to study the effectiveness of treatment with methotrexate and cyclosporine after bone marrow transplantation to provide protection against acute graft-versus-host disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of a combination of methotrexate and cyclosporine, administered after grafting, to prevent the development of acute graft versus host disease (GVHD) in patients undergoing allogeneic bone marrow transplantation.

OUTLINE: Patients receive methotrexate IV on days 1,3,6, and 11. Patients also receive cyclosporine IV twice a day until the patient is eating, then it is administered orally twice a day. Cyclosporine begins on day -1 and continues until day 180. The dose is reduced beginning on day 50.

PROJECTED ACCRUAL: Accrual will continue until further notice.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Ongoing bone marrow transplantation from HLA-matched siblings or HLA non-identical family members or unrelated donor

PATIENT CHARACTERISTICS: Age: Any age Performance status: Not specified Life expectancy: Not severely limited by disease other than leukemia Hematopoietic: Not specified Hepatic: No severe hepatic disease Renal: No history of hemorrhagic cystitis No renal disease Cardiovascular No symptomatic cardiac disease Other: No contraindication to the use of cyclosporine or methotrexate

PRIOR CONCURRENT THERAPY: No concurrent experimental treatment on other GVHD prophylaxis studies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1986-05; Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer F. Storb, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States